CLINICAL TRIAL: NCT07322224
Title: A Multi-Modal Longevity Protocol Integrating Lifestyle, Supplements, and Autologous Pro-Regenerative Cell-Conditioned Media: A Pilot Study
Brief Title: Multi-Modal Longevity Protocol Including Autologous Cell-Free Conditioned Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BlueBird Age Reversal SA (Industry)
Collaborators: xLongevity (Unknown); Wellbeing International Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BB-ART3-2024-PILOT
Record Dates: First submitted 2025-12-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Biological Aging; Healthy Aging; Longevity
Keywords: Epigenetic age; Phenotypic age; Autologous conditioned media; Longevity protocol; Supplements; Lifestyle

STUDY DESIGN:
Intervention Model Description: Single-arm exploratory study in which all participants received the same multi-modal longevity protocol, including lifestyle optimisation, nutritional supplementation, and autologous cell-free conditioned media (APRC-CM). No comparator group was included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Longevity Protocol Arm (Experimental): Participants received a structured, multi-modal longevity protocol consisting of lifestyle optimization, nutritional supplementation, and autologous cell-free conditioned media (APRC-CM) prepared individually from peripheral blood-derived pro-regenerative cells. All participants received the same intervention schedule over a 17-week period.
  Interventions: Behavioral: Multi-Modal Longevity Protocol

INTERVENTIONS:
Behavioral: Multi-Modal Longevity Protocol — The intervention consisted of a structured, multi-modal longevity program that included lifestyle optimization (nutrition, physical activity, and sleep routines), nutritional supplementation, and autologous cell-free conditioned media (APRC-CM). APRC-CM was prepared individually for each participant from peripheral blood-derived pro-regenerative cells and administered as part of a physiologic, minimal-risk exploratory protocol.

SUMMARY:
This pilot study evaluated a multi-modal longevity protocol combining lifestyle optimisation, nutritional supplementation, and autologous cell-free conditioned media derived from peripheral blood-derived pro-regenerative cells (APRC-CM). Fourteen healthy adult participants completed a 17-week programme including baseline and post-intervention biomarker assessments. The primary objective was to characterise changes in biological age using DNA methylation-based epigenetic clocks, PhenoAge and other physiological and biochemical markers.

DETAILED DESCRIPTION:
This exploratory study investigated the biological effects of a structured, multi-modal longevity programme that included lifestyle optimisation (nutrition, exercise, sleep routines), nutritional supplementation, and autologous cell-free conditioned media (APRC-CM). APRC-CM was prepared individually for each participant from peripheral blood-derived pro-regenerative cells cultured ex vivo to produce a pro-regenerative secretome containing soluble factors and extracellular vesicles.

Participants underwent biomarker assessments at baseline and at week 17. Outcomes included measurements of epigenetic biological age, phenotypic age, inflammatory markers, metabolic markers, and other laboratory and physiological variables. The study was conducted in healthy adults and designed as a minimal-risk physiological investigation.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 years or older
* Generally good overall health as assessed by the study team
* Able and willing to provide written informed consent
* Willing to participate in all components of the study protocol, including lifestyle optimisation, nutritional supplementation, blood collection, and scheduled follow-up visits
* Able to comply with study procedures for the duration of the intervention and assessments

Exclusion Criteria:

* Presence of a major medical condition that, in the opinion of the investigators, could affect participation or safety
* Any condition requiring hospitalization or emergency medical intervention within the past 12 months
* Receipt of anti-aging or longevity treatments within the past six months (e.g., intravenous therapies, regenerative or cellular treatments, structured age-reversal programmes)
* Active infectious disease at enrolment
* Pregnancy or breastfeeding
* Use of systemic immunomodulatory, cytotoxic, or investigational treatments in the prior 3 months
* Any condition or circumstance that, in the judgement of the investigators, may interfere with study participation or data integrity

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Epigenetic Biological Age | Baseline and Week 17
  Biological age calculated from DNA methylation profiles using validated epigenetic clock algorithms.

SECONDARY OUTCOMES:
Change in Phenotypic Age | Baseline and Week 17
  Phenotypic age calculated from clinical biomarkers using published phenotypic age algorithms.

OTHER OUTCOMES:
Incidence of Adverse Events | From baseline to Week 17
  Monitoring of any self-reported or observed adverse events throughout the study period. Events were recorded and assessed descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Ortega, MD, Principal Investigator — Wellbeing International Foundation
Locations (1):
- Wellbeing International Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset includes biological, clinical, and demographic information that may be potentially identifiable, and no data-sharing agreements or infrastructure were established for this pilot study.